CLINICAL TRIAL: NCT06960850
Title: A Randomized Controlled Trial on the Effect of Oral Propranolol on Induction-Delivery Interval in Women Undergoing Oxytocin Induction of Labour in Abakaliki
Brief Title: Effects of Oral Propranolol on Induction-Delivery Interval During Induction of Labour With Oxytocin
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Federal Teaching Hospital Abakaliki (Other Government)
Responsible Party: Principal Investigator, Assumpta Nnenna Nweke, Principal Investigator, Federal Teaching Hospital Abakaliki
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: AE-FUTHA/REC/VOL3/2024/409
Record Dates: First submitted 2025-04-29; First posted 2025-05-07 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-04

CONDITIONS: Propranolol; Labour Induction
Keywords: Propanolol; Induction-Delivery; Oxytocin; Labour Induction
MeSH Terms: interventions — Propranolol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Propranolol (Experimental): A set of 154 numbers will receive oxytocin and propranolol once or twice 6 hours apart. The first dose will be from 10 minutes before commencement of oxytocin titration and the second dose will be 6 hours from the first dose if delivery has not taken place.
  Interventions: Drug: Propranolol
- Placebo (Placebo Comparator): A set of 154 numbers will receive oxytocin and placebo once or twice 6 hours apart. The first dose will be from 10 minutes before commencement of oxytocin titration and the second dose will be 6 hours from the first dose if delivery has not taken place.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Propranolol — A set of 154 numbers will receive oxytocin and propranolol once or twice 6 hours apart. the first dose will be from 10 minutes before commencement of oxytocin titration and the second dose will be 6 hours from the first dose if delivery has not taken place.
  Arms: Propranolol
Other: Placebo — A set of 154 numbers will receive oxytocin and placebo once or twice 6 hours apart. the first dose will be from 10 minutes before commencement of oxytocin titration and the second dose will be 6 hours from the first dose if delivery has not taken place.
  Arms: Placebo

SUMMARY:
Prolonged pregnancy could lead to perinatal and maternal complications. Oxytocin has been wildly used for induction of labour, but prolonged labour continued to occur with its attendant sequelae. Propranolol, a non-selective B-adrenergic inhibitor has been found to facilitate labour progress in some studies, by the blockade of the effects of catecholamines on the uterus though there are conflicting reports, with the only meta-analysis inconclusive due to few studies used; hence, the need to further study its role in induction of labour. The aim of this study is to assess the role of oral Propranolol in decreasing the induction-delivery with oxytocin

DETAILED DESCRIPTION:
Background: Prolonged pregnancy could lead to perinatal and maternal complications. To prevent this, induction of labour becomes necessary. Conventionally, oxytocin has been wildly used for induction of labour, but prolonged labour continued to occur with its attendant sequelae. Propranolol, a non-selective B-adrenergic inhibitor has been found to facilitate labour progress in some studies, by the blockade of the effects of catecholamines on the uterus though there are conflicting reports, with the only meta-analysis inconclusive due to few studies used; hence, the need to further study its role in induction of labour.

Aim: The aim of this study is to assess the role of oral Propranolol in decreasing the induction-delivery with oxytocin.

Methodology: This will be double-blind, superiority randomised controlled trial involving pregnant women at term who meet the inclusion criteria and consent to the study over a six-month period. The participants will be randomised by means of computer-generated numbers from a pool of 308 participants. A set of 154 numbers will receive oxytocin + propranolol once/twice 6 hours apart, starting from 10 minutes before commencement of oxytocin titration; while the other set of 154 numbers would be given oxytocin + placebo once/twice 6 hours apart, starting from 10 minutes before commencement of oxytocin titration.Labour will be monitored with the labour care guide.

ELIGIBILITY:
Inclusion Criteria:

* singleton foetus
* cephalic presentation at term

Exclusion Criteria:

* Patients on beta blockers
* Contraindications to labour or vaginal delivery
* Multiple gestations
* Preterm labour
* Chorioamnionitis
* Known fetal anomalies
* Bronchial asthma
* Abnormal fetal presentation.
* Antepartum haemorrhage.
* Lung disease
* Previous uterine scar or surgery.
* Foetal heart irregularity

Ages: 15 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 308 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Mean duration of first, second and third stage of labour | 24 hours
  this is to assess the mean duration of the first, second and third stages of labour

CONTACTS AND LOCATIONS:
Locations (1):
- Alex Ekwueme Federal University Teaching Hospital, Abakaliki, Ebonyi State, Nigeria

IPD SHARING:
Plan to Share IPD: No